CLINICAL TRIAL: NCT00478868
Title: Modic Changes and Associated Features in Southern European Chronic Low Back Pain Patients
Acronym: MODIC
Status: Completed | Type: Observational
Sponsor: Kovacs Foundation (Other)
Responsible Party: Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation
Other Study IDs: FK-R-15
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Low Back Pain
Keywords: MODIC changes; chronic low back pain; magnetic resonance imaging (MRI); vertebrae; intervertebral disc
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To assess: a) The prevalence of Modic changes and other findings on lumbar magnetic resonance imaging (MRI), among Spanish adult chronic LBP patients, b) Patient characteristics and radiological findings associated with Modic changes.

DETAILED DESCRIPTION:
Ten radiologists from six hospitals across six cities in Spain, consecutively recruited 487 adult patients (263 women and 224 men) in whom lumbar MRI had been prescribed for low back pain lasting ≥ 3 months. Patients' characteristics and imaging findings were assessed through previously validated instruments. A multivariate logistic regression model was developed to assess the features associated with Modic changes.

Outcome measures were: Gender, age, body mass index (BMI), life time smoking exposure, degree of physical activity, and image features (disk degeneration, type and extension of Modic changes, disk contour, annular tears, spinal stenosis and spondylolisthesis).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 35 and 50 years of age having a diagnosis of chronic low back pain (of 3 or more months' duration, and including sciatica and lumbar cytalgia), who get a prescription for an MRI.

Exclusion Criteria:

* Racial characteristics suggesting a non-Spanish origin; central nervous system pathology (with or without treatment);
* Diagnosis or suspicion of systemic disease (inflammatory disease such as rheumatoid arthritis, or infections).

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients seen for chronic low back pain at the hospitals of the Spanish National Health Service.
Sampling Method: Non-Probability Sample
Enrollment: 487 (Actual)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Modic change | Upon assessment
  Modic change type, extension and volume

SECONDARY OUTCOMES:
Patients' characteristics | Upon assessment
  Gender, age, body mass index (BMI), life time smoking exposure, and degree of physical activity
Image features | Upon assessment
  Disk degeneration, type and extension of Modic changes, disk contour, annular tears, spinal stenosis and spondylolisthesis

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, Spain; Carlos Campillo, MD, Principal Investigator — IbSalut, Palma de Mallorca, Spain
Locations (1):
- Kovacs Foundation, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Background] Modic MT, Steinberg PM, Ross JS, Masaryk TJ, Carter JR. Degenerative disk disease: assessment of changes in vertebral body marrow with MR imaging. Radiology. 1988 Jan;166(1 Pt 1):193-9. doi: 10.1148/radiology.166.1.3336678.
- [Background] Toyone T, Takahashi K, Kitahara H, Yamagata M, Murakami M, Moriya H. Vertebral bone-marrow changes in degenerative lumbar disc disease. An MRI study of 74 patients with low back pain. J Bone Joint Surg Br. 1994 Sep;76(5):757-64. PMID 8083266
- [Background] Stirling A, Worthington T, Rafiq M, Lambert PA, Elliott TS. Association between sciatica and Propionibacterium acnes. Lancet. 2001 Jun 23;357(9273):2024-5. doi: 10.1016/S0140-6736(00)05109-6. No abstract available. PMID 11438138